CLINICAL TRIAL: NCT06447207
Title: Social Prescription for Loneliness in Community-based Group Exercise Classes for People With Parkinson Disease
Brief Title: Occupational Therapy Led Social Prescription for People With Parkinson Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5561; AOTFIR24Swink (Other: American Occupational Therapy Foundation)
Record Dates: First submitted 2024-05-21; First posted 2024-06-07 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Loneliness; Social Prescription
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: single group trial of occupational therapy led social prescription program for people with Parkinson disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occupational Therapy Led Social Prescription (Experimental): (1) A baseline occupational therapy assessment including a social prescription, (2) Six monthly occupational therapy follow-up sessions focused on behavior-change techniques to encourage participation in the social prescription, and include: review of the social prescription, self-monitoring strategies, facilitators review, barriers review, problem-solving, provision of feedback, action planning, and rating confidence with the action plan, and (3) Post Occupational Therapy Assessment
  Interventions: Behavioral: Occupational Therapy Led Social Prescription

INTERVENTIONS:
Behavioral: Occupational Therapy Led Social Prescription — The intervention includes encouragement to participate in the co-designed social prescription with 6 monthly sessions with an occupational therapist or occupational therapy doctoral student.

SUMMARY:
Loneliness is an epidemic that the U.S. Surgeon General implored must be addressed by society as a whole. Increased loneliness (i.e., distressing feelings of isolation) in people with Parkinson's disease (PD) has a pervasive impact and is associated with worsened motor and non-motor symptoms, and quality of life. The investigators expect that individuals participating socially in the community would experience less loneliness. However, for individuals with PD participating in community-based group exercise programs, the investigators have found that over one third still report being lonely. Therefore, an evidence-based program needs to be added to address a significant problem of loneliness for people with PD-and occupational therapy is the leading discipline to add the intervention because social participation is one of eight occupations that an occupational therapist is focused on optimizing. The chief executive officer at the Parkinson Association of the Rockies (PAR), members of the Colorado State University Occupational Therapy Department, and members of the University of Colorado's Parkinson's Exercise Research Consortium have teamed up to address pervasive loneliness.

Social prescription is a prime evidence-based intervention to add to existing PD community-based exercise classes because it has been shown to reduce loneliness. For this project, the investigators detect participants in the 'lonely' range through a standardized assessment. The investigators will work with PAR staff who will refer individuals identifying as 'lonely' to an occupational therapist, who will complete an individualized occupational profile and write the appropriate social prescription from 11 different interventions (examples include: intergenerational intervention, animal companions, physical activity, occupational therapy) from established community resources recommended for social prescription. The proposed project is designed with three primary goals: (1) determine the reach of the social prescription program, (2) evaluate the effectiveness of the program at one site, and (3) determine implementation strategies for scalability.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative condition with no known cure. Current evidence-based practice focuses on slowing disease progression, reducing negative impacts of motor and non-motor symptoms, and improving quality of life. While approaches such as exercise, medications, and surgery are used to reduce impacts of PD symptoms, there is a gap in how to address loneliness, which is a significant factor associated with poor quality of life for people with PD. Loneliness is a vast problem in the United States, the Surgeon General released a 2023 report imploring a societal focus on addressing loneliness (i.e., distressing feelings of isolation)-and people with PD have an even higher prevalence of loneliness than the general population. Occupational therapists play a key role in addressing the loneliness epidemic for people with PD. Social participation is one of eight categories of occupation elucidated in the Occupational Therapy (OT) Practice Framework. Yet, limited OT guidelines exist on how to address the occupation of social participation. According to the 2022 OT Clinical Practice Guidelines for people with PD, moderate evidence exists for community-based group activity. Considering OT as a discipline focused on using occupation both as a means (training using social participation), and as an ends (reduction of loneliness), investigators should be on the forefront of evidence-based practice to address loneliness. Group format, community-based exercise is one approach with potential for addressing loneliness. Parkinson Association of the Rockies (PAR) offers 70+ weekly community-based group exercise classes in Colorado and surrounding states. For over two years, the investigators have been partnering with PAR to collect outcomes data of PAR exercise class participants in areas of psychosocial outcomes (e.g., loneliness), mobility, and quality of life. Interestingly, over one third of individuals with PD who are participating in the PAR group exercise classes self-report to be in the 'lonely' range (3-item UCLA Loneliness Scale [UTILS] score =5/9). After reviewing evidence-informed strategies to address loneliness, the investigators found a clear method already developed-social prescription. Social prescription offers a method to improve loneliness through further community connection in an individualized, meaningful way.

Evidence-based Practice to Address Loneliness

The process of social prescription is standardized, requiring identification into the program by a health professional or community member (e.g., PAR staff), evaluation with a coordinator (e.g., OT), and partnerships with local organizations (e.g., PAR). The investigators developed a preliminary resource manual to identify resources within each of the 11 interventions recommended within social prescription (e.g., intergenerational intervention, animal companions, physical activity, occupational therapy), and use an occupational profile to identify the individualized target area for each participant. The approach will follow the Grol & Wensing Implementation Process model in which the investigators have already completed Steps 1-3 (identifying the topic for change, analysis of sample/site, selection of strategies to address change). Now in steps 4&5 of the model, the investigators will implement social prescription with one organization, and then evaluate to adapt prior to scaling up to multiple organizations, with the following two aims:

Aim 1. Determine the reach of OT-led social prescription for people with Parkinson's disease using a single-site pilot trial.

Aim 2. Evaluate the OT-led social prescription for people with Parkinson's disease for a signal of effectiveness using a single-site pilot trial.

Aim 3. Determine implementation strategies to facilitate scalability of OT-led social prescription beyond the single-site and Colorado community.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Have a diagnosis of Parkinson Disease
* Have participated in at least one exercise class or support group in the last year
* Scored ≥5/9 on the UCLA 3-item Loneliness Scale during pre-screening
* Agree to participate in a 6-month program including a social prescription and six visits with an occupational therapist or occupational therapy doctoral student

Exclusion Criteria:

* Have ever been diagnosed with dementia
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The Three-Item Loneliness Scale | baseline, pre-intervention and immediately after the intervention
  The Three-Item Loneliness Scale is an assessment of loneliness scored 3-9 with higher scores indicating greater (worse) loneliness.

SECONDARY OUTCOMES:
Study Reach | during the intervention
  (1) % of participants screened for loneliness by PAR assessors in each class/total people in the class, (2) % eligible/total people screened, (3) % who enroll in OT-led social prescription/total people eligible, (4) # OT follow-up sessions completed (out of 6 total) on average for people who enrolled
Social Participation and Social Activities | baseline, pre-intervention and immediately after the intervention
  Activity Card Sort Version 2 scores range from 0-100 with higher scores indicating greater retention of social roles and activities since diagnosis.
Health-related Quality of Life with Social Satisfaction Focus | baseline, pre-intervention and immediately after the intervention
  The Satisfaction with Social Roles and Activities Short Form scores range from 8-40 with higher scores indicating greater satisfaction with social roles and activities.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Swink, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No